CLINICAL TRIAL: NCT05027243
Title: Outcomes of Bilateral Temporomandibular Joint Arthroscopy and the Role of a Second Intervention - Timings and Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Portugues da Face (Other)
Responsible Party: Principal Investigator, David Faustino Ângelo, Clinical Director, Instituto Portugues da Face
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMJARTHRO
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Bilateral Temporomandibular Joint Disorder
Keywords: Temporomandibular joint; TMJ arthroscopy; TMJ surgery
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: Prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bilateral temporomandibular joint arthroscopy (Experimental)
  Interventions: Procedure: bilateral temporomandibular joint arthroscopy; Drug: Xeomin® (Merz)

INTERVENTIONS:
Procedure: bilateral temporomandibular joint arthroscopy — The TMJ arthroscopy was performed with a 1.9-mm arthroscope including a video system, with a 2.8-mm outer protective cannula. Briefly, for TMJ arthroscopy level 1, the authors used the classic puncture with an entry point 10 mm anterior and 2 mm below the Holmlund-Hellsing (H-H) line. A second puncture with a 21-G needle was performed 30 mm anterior and 7 mm below the H-H line to wash the joint with 250-300 ml Ringer solution. After washing the joint, 1.5-2 cc of hyaluronic acid was injected into it. For level 2 TMJ arthroscopy, the second puncture was substituted by a 2.8-mm outer protective cannula with a sharp trocar until the joint was reached. The 2.8-mm cannula was used for (1) intra-articular coblation and/or (2) intrasynovial medication. Antibiotic and non-steroidal anti-inflammatory drugs were routinely prescribed. Patients were instructed to follow a soft diet for 3 days after surgery and 5 physiotherapy and 3 speech therapy exercise sessions after intervention.
Drug: Xeomin® (Merz) — For tenderness grade 2, 155U of Incobotulinum toxin A was injected in the masticatory muscles and for tenderness grade 3 195U of Incobotulinum toxin A was injected. The authors used Xeomin® (Merz) in all patients.

SUMMARY:
Temporomandibular joint (TMJ) arthroscopy has been used successfully for intra-articular disorders. Until now, limited studies are available regarding the clinical evidence of bilateral TMJ arthroscopy for Dimitroulis 2-3. This prospective study investigated the efficacy of TMJ arthroscopy in patients with bilateral disorders, and also the need for a posterior surgery.

DETAILED DESCRIPTION:
Temporomandibular joint (TMJ) arthroscopy has been used successfully for intra-articular disorders. It was first introduced by Onishi at 1975, as a pioneering technique to treat painful joints and has been associated with a reduction in the number of open joints surgeries. This minimally invasive technique allows observation of the TMJ upper compartment tissues, and sometimes the lower compartment. Moreover, this intervention allows joint lysis and lavage (level 1 arthroscopy) and intra-articular surgical procedures (level 2-3 arthroscopy).

Recent studies updated that TMJ arthroscopy promotes a reduction in pain and inflammatory process and restoring the mandibular function with low morbidity. Moreover, TMJ arthroscopy seems to be also long-term effective for relieving TMJ symptoms. Until now, limited studies are available regarding the clinical evidence of bilateral TMJ arthroscopy for Dimitroulis 2-3. This prospective study investigated the efficacy of TMJ arthroscopy in patients with bilateral disorders, and also the need for a posterior surgery.

ELIGIBILITY:
Inclusion Criteria:

* age >16 years;
* clinical diagnosis of bilateral intra-articular disorder;
* clinical criteria for bilateral TMJ arthroscopy;
* magnetic resonance imaging (MRI) assessing the intra-articular derangement

Exclusion Criteria:

* The exclusion criteria included any history of previous TMJ surgical intervention or any facial trauma within the last 4 weeks prior the study.
* Severe medical problems or mental illness, and pregnancy were also exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Pain (Visual Analogue Scale (0,10) | Pre-surgery
  VAS, 0-10, with 0 being no pain and 10 having maximum unbearable pain
Pain (Visual Analogue Scale (0,10) | Through study completion, an average of 2.5 years
  VAS, 0-10, with 0 being no pain and 10 having maximum unbearable pain

SECONDARY OUTCOMES:
Maximum mouth opening (MMO, mm) | Pre-surgery
  Mouth opening measured with a ruler (mm)
Maximum mouth opening (MMO, mm) | Through study completion, an average of 2.5 years
  Mouth opening measured with a ruler (mm)
Muscle tenderness (0-3 scale) | Pre-surgery
  0-3, corresponding to a muscle tenderness scale in masseter and temporalis muscle (0-whithout muscle tenderness, 3 - maximum muscle tenderness)
Muscle tenderness (0-3 scale) | Through study completion, an average of 2.5 years
  0-3, corresponding to a muscle tenderness scale in masseter and temporalis muscle (0-whithout muscle tenderness, 3 - maximum muscle tenderness)

CONTACTS AND LOCATIONS:
Overall Officials: David Ângelo, MD, PhD, Principal Investigator — Instituto Português da Face

IPD SHARING:
Plan to Share IPD: No